CLINICAL TRIAL: NCT04980235
Title: Evaluation of Levator Ani Muscle Injury in Primiparous Women at One and Six Weeks Postpartum Using 4D Transperineal Ultrasound: Comparative Cohort Study
Brief Title: Evaluation of Levator Ani Muscle Injury in Primiparous
Acronym: ULTRASOUND
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mervit Sersy, Assistant professor, Alexandria University
Other Study IDs: 0305043
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Pelvic Floor Disorders
Keywords: levator hiatus
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transperineal 3D ultrasound — All ultrasound volumes were acquired 7days after delivery and another examination 6weeks post-delivery by one experienced sonographers using a GEVoluson p8 (GE Healthcare) equipped with a 4-8-MHz curved array 3Dultrasound transducer

SUMMARY:
pelvic floor muscles play an important role in supporting the pelvic organs. Vaginal birth leads to defects in pelvic muscles and hence subsequent pelvic organ prolapse and urinary and fecal incontinence can occur . Transperineal ultrasonography study pelvic floor pathology with minimal discomfort to the patient and lower cost than magnetic resonance imaging.

DETAILED DESCRIPTION:
355 eligible Egyptian women had been enrolled Maternal Medical, surgical and obstetrical history was obtained. Demographic data (maternal age, maternal body mass index, duration of second stage labor, episiotomy, maternal injuries, neonatal birth weight, and neonatal head circumference were obtained. A modified questionnaire on symptoms of pelvic floor dysfunction was filled by the patients in both visits. vaginal examination with the women to detect any pelvic organ prolapse (quantified according to POP-Q classification system.

All ultrasound volumes were acquired 7days after delivery and another examination 6weeks post-delivery by one experienced sonographers using a GE Voluson p8 (GE Healthcare) equipped with a 4-8-MHz curved array 3D/4D ultrasound transducer. After emptying the bladder, ultrasound was done while the patient in the supine position. The probe was covered with clean glove adjusted and wrapped with an adhesive tape to make it firmly contacted to the probe and then placed on the perineum in the sagittal plane. The field of view angle was set to a maximum of 70° in the sagittal plane and the volume acquisition angle to 85° in the axial plane. Two 3D volumes (one with the patient at rest and one during Valsalva maneuver) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Primipara who had singleton fetus with cephalic presentation were recruited during their first post-partum visit ,1week post-delivery.

Exclusion Criteria:

Multi para, Multifetal pregnancy, congenital anomalies of the genital tract past history of pelvic floor surgery or trauma or inability to come for follow up after 6weeks

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was performed at Shatby maternity university hospital in Alexandria where 12000 deliveries per year are achieved . Over a 4-months period (February-June 2021.
  355 eligible Egyptian women
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
1. maximum diameters of the levator hiatus , pubovisceral muscle thickness Levator avulsion . | 6weeks
  Measurements were performed in the axial plane at the level of 'minimal hiatal dimensions'

CONTACTS AND LOCATIONS:
Overall Officials: Mervat AM Elsersy, MD, Principal Investigator — Assistant professor
Locations (1):
- Shatby Maternity University Hospital, Alexandria, El-Khartoum Square, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie result
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication).
Access Criteria: all individuals in the same institution
URL: http://www.med.alexu.edu.eg